CLINICAL TRIAL: NCT00957996
Title: A Phase 3, Open-Label, Randomized Study of the Antiviral Activity, Safety, and Tolerability of Intravenous Peramivir in Hospitalized Subjects With Confirmed or Suspected Influenza Infection
Brief Title: Safety Study of IV Peramivir in Hospitalized Subjects With Confirmed or Suspected Influenza
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: BioCryst Pharmaceuticals (Industry)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BCX1812-303; HHS 0100200700032C (Other Grant/Funding Number: HHS-BARDA)
Record Dates: First submitted 2009-08-12; First posted 2009-08-13 (Estimated); Results first posted 2015-02-12 (Estimated); Last update posted 2015-02-12 (Estimated); Status verified 2015-01

CONDITIONS: Seasonal Influenza; Cough; Sore Throat; Nasal Congestion; Myalgia; Headache; Fatigue
Keywords: influenza; hospitalized; flu; antiviral
MeSH Terms: conditions — Cough; Pharyngitis; Nasal Obstruction; Myalgia; Headache; Fatigue; Influenza, Human | interventions — peramivir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Peramivir 300 mg (Experimental): Peramivir 300 mg twice daily
  Interventions: Drug: Peramivir
- Peramivir 600 mg (Experimental): Peramivir 600 mg once daily
  Interventions: Drug: Peramivir

INTERVENTIONS:
Drug: Peramivir — 300 mg twice daily
  Arms: Peramivir 300 mg
Drug: Peramivir — 600 mg once daily
  Arms: Peramivir 600 mg

SUMMARY:
This is a Phase 3, open-label, randomized study of the antiviral activity, safety, and tolerability of intravenous Peramivir in hospitalized subjects with confirmed or suspected influenza infection.

ELIGIBILITY:
Inclusion Criteria:

* Male and non-pregnant female subjects 6 years of age or older.
* Able to provide written informed consent, or for whom written consent may be provided by a parent guardian or legally authorized representative, unless consent provided by a parent, guardian or legally authorized representative is not consistent with applicable local or ethical procedures, directives and /or guidelines.
* Presence of clinical signs and/or symptoms consistent with an acute illness compatible with influenza infection; a measured temperature of ≥ 38.0°C (100.4°F) oral, or ≥ 38.6°C (101.4°F) rectal or tympanic and recent onset of at least one of the following: rhinorrhea or nasal congestion, sore throat or cough. Measured temperature can include fever meeting the above criteria as reported by the subject or their parent, guardian or legally authorized representative in the 24 hours prior to Screening. The requirement for fever is waived for any subject with influenza infection already confirmed by laboratory tests (including Rapid Antigen Tests).
* Confirmation of influenza A or B infection in the local community by one of the following means:
* the institution's local laboratory,
* the local public health system
* the national public health system
* a laboratory of a recognized national or multinational influenza surveillance scheme.
* Severity of illness requiring or anticipated to require in-hospital care.

Exclusion Criteria:

* Subjects who have been hospitalized for greater than 24 hours (not including time spent in the emergency department).Blood platelet count of < 20 x 109/L.
* Serum bilirubin > 6 mg/dL at time of Screening evaluation.
* Serum ALT or AST > 5 X upper limit of normal at time of Screening evaluation.
* Serum creatinine > 5.0 mg/dL at time of Screening evaluation.
* Subjects who require peritoneal dialysis or hemofiltration.
* Altered neurologic status as defined by a Glasgow Coma Score of ≤ 9, unless medically induced.
* Females who are pregnant (positive urine or serum pregnancy test at Screening evaluation) or breastfeeding.
* Actively undergoing systemic chemotherapy or radiotherapy treatment for a malignancy. (Subjects who have completed treatment 30 days prior to enrollment are allowed to enroll in the study. Hormone treatment for cancer is also acceptable).
* Prior hematopoietic stem cell transplantation or solid organ transplant during the previous 4 months.
* HIV infection with a known CD4 count < 200 cells/ mm3 unless on a stable highly active antiretroviral (HAART) regimen for at least 6 months.
* Presence of a preexisting chronic infection that is undergoing or requiring medical therapy (eg, tuberculosis). (Subjects with chronic osteomyelitis or hepatitis B or C not requiring treatment are not excluded).
* Presence of any preexisting illness that, in the opinion of the Investigator, would place the subject at an unreasonably increased risk through participation in this study.
* Participation as a subject in any study of an experimental treatment for any condition within the 30 days prior to the time of the Screening evaluation.
* Subjects diagnosed with cystic fibrosis.
* Subjects with confirmed clinical evidence of acute non-influenzal infection at the time of Screening.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2009-10; Primary Completion 2010-10 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (110):
- United States (79):
  - Dothan, Alabama
  - Mobile, Alabama
  - Jonesboro, Arkansas
  - Little Rock, Arkansas
  - Fountain Valley, California
  - Harbor City, California
  - La Mesa, California
  - Long Beach, California
  - Los Angeles, California
  - Modesto, California
  - Oceanside, California
  - Orange, California
  - Palo Alto, California
  - Sacramento, California
  - San Diego, California
  - San Francisco, California
  - San Jose, California
  - Denver, Colorado
  - Wheat Ridge, Colorado
  - Washington D.C., District of Columbia
  - Brandon, Florida
  - Fort Lauderdale, Florida
  - Gainsville, Florida
  - Ocoee, Florida
  - Orlando, Florida
  - West Palm Beach, Florida
  - Columbus, Georgia
  - Decatur, Georgia
  - Honolulu, Hawaii
  - Idaho Falls, Idaho
  - Chicago, Illinois
  - Rock Island, Illinois
  - Springfield, Illinois
  - Indianapolis, Indiana
  - South Bend, Indiana
  - Topeka, Kansas
  - Hazard, Kentucky
  - Natchitoches, Louisiana
  - Shreveport, Louisiana
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Detroit, Michigan
  - Royal Oak, Michigan
  - Troy, Michigan
  - Minneapolis, Minnesota
  - St Louis, Missouri
  - Butte, Montana
  - Omaha, Nebraska
  - Englewood, New Jersey
  - Hackensack, New Jersey
  - Neptune City, New Jersey
  - New Brunswick, New Jersey
  - Somers Point, New Jersey
  - Albuquerque, New Mexico
  - Albany, New York
  - Brooklyn, New York
  - Buffalo, New York
  - Jamaica, New York
  - New York, New York
  - The Bronx, New York
  - Valhalla, New York
  - Akron, Ohio
  - Cleveland, Ohio
  - Lima, Ohio
  - Toledo, Ohio
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Providence, Rhode Island
  - Charleston, South Carolina
  - Sioux Falls, South Dakota
  - Houston, Texas
  - San Antonio, Texas
  - Tomball, Texas
  - Salt Lake City, Utah
  - Norfolk, Virginia
  - Salem, Virginia
  - Bellevue, Washington
  - Seattle, Washington
  - Milwaukee, Wisconsin
- Australia (6):
  - Brisbane, Queensland
  - Cairns, Queensland
  - Southport, Queensland
  - Clayton, Victoria
  - Melbourne, Victoria
  - Parkville, Victoria
- Canada (13):
  - Kelowna, British Columbia
  - Winnipeg, Manitoba
  - Hamilton, Ontario
  - Kingston, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
  - Chicoutimi, Quebec
  - Montreal, Quebec
  - Sainte-Foy, Quebec
  - Sherbrooke, Quebec
  - Trois-Rivières, Quebec
  - Saskatoon, Saskatchewan
  - Edmonton
- Mexico (7):
  - Aguascalientes, Aguascalientes
  - Guadalajara, Jalisco
  - Zapopan, Jalisco
  - Distrito Federal, Mexico City
  - Monterrey, Nuevo León
  - San Luis Potosí City, San Luis Potosí
  - Durango
- New Zealand (4):
  - Auckland, Wellington Region
  - Christchurch
  - Hamilton
  - Tauranga
- San Juan, Puerto Rico

REFERENCES:
- [Derived] Ison MG, Fraiz J, Heller B, Jauregui L, Mills G, O'Riordan W, O'Neil B, Playford EG, Rolf JD, Sada-Diaz E, Elder J, Collis P, Hernandez JE, Sheridan WP. Intravenous peramivir for treatment of influenza in hospitalized patients. Antivir Ther. 2014;19(4):349-61. doi: 10.3851/IMP2680. Epub 2013 Aug 28. PMID 23985625

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Peramivir 300 mg | Peramivir 600 mg
Started | 117 | 117
Completed | 91 | 89
Not Completed | 26 | 28
Not completed — Death | 4 | 10
Not completed — Lost to Follow-up | 4 | 7
Not completed — Withdrawal by Subject | 9 | 2
Not completed — Adverse Event | 2 | 1
Not completed — Physician Decision | 1 | 1
Not completed — Influenza-related complication | 0 | 1
Not completed — Missing | 1 | 0
Not completed — Noncompliance; Protocol Deviations | 5 | 6

BASELINE CHARACTERISTICS:
Population: The Intent-to-Treat (ITT) population included all randomized subjects.
Groups:
- Peramivir 300mg: 300 mg twice daily
  Peramivir: 300 mg twice daily
- Peramivir 600mg: 600 mg once daily
  Peramivir: 600 mg once daily
- Total: Total of all reporting groups
Arm/Group | Peramivir 300mg | Peramivir 600mg | Total
Number analyzed (Participants) | 117 | 117 | 234
Age, Continuous [Mean (Full Range); unit: years] | 48.3 [14 to 93] | 48.4 [15 to 92] | 48.3 [14 to 93]
Age, Customized [Number; unit: participants]
  Children 6-11 years | 0 | 0 | 0
  Adolescents 12-17 years | 3 | 1 | 4
  Adults 18-24 years | 4 | 8 | 12
  Adults 25-34 years | 17 | 19 | 36
  Adults 35-44 years | 29 | 18 | 47
  Adults 45-54 years | 26 | 29 | 55
  Adults 55-64 years | 18 | 27 | 45
  Adults 65-74 years | 11 | 10 | 21
  Adults ≥75 years | 9 | 5 | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 65 | 139
  Male | 43 | 52 | 95
Race/Ethnicity, Customized [Number; unit: participants]
  White | 78 | 84 | 162
  Black, of African Heritage or African American | 16 | 13 | 29
  Other | 15 | 11 | 26
  Asian | 5 | 5 | 10
  American Indian or Alaska Native | 3 | 1 | 4
  Native Hawaiian or other Pacific Islander | 0 | 3 | 3
Body mass index (BMI) [Mean (Full Range); unit: kg/m^2] | 32 [17 to 70] | 31 [18 to 59] | 31 [17 to 70]
Smoking status [Number; unit: participants]
  Current smoker | 43 | 45 | 88
  Not current smoker | 73 | 72 | 145
  Missing | 1 | 0 | 1
Influenza vaccination status [Number; unit: participants] — Subjects may have had more than one vaccination.
  participants
    Not vaccinated this year | 74 | 81 | 155
    Vaccinated this year | 41 | 36 | 77
    Missing | 2 | 0 | 2
Number of subjects with ICU admission at Baseline [Number; unit: participants] | 18 | 21 | 39
APACHE II Score [Mean (Standard Deviation); unit: units on a scale] — Acute physiology and chronic health evaluation (APACHE) Score was captured only for the first ICU admission. The APACHE II Score ranges from 0 to 71 with higher scores indicating greater disease severity and a higher risk of death.
  units on a scale | 14 (7.5) | 17 (5.4) | 15 (6.6)
Chest X-ray at Screening [Number; unit: participants]
  Normal | 82 | 86 | 168
  Abnormal | 31 | 28 | 59
  Missing | 4 | 3 | 7
Duration of illness [Number; unit: participants]
  ≤48 hours | 18 | 16 | 34
  >48 hours | 99 | 101 | 200
Hemisphere of enrollment [Number; unit: participants]
  Northern Hemisphere 09-10 | 107 | 108 | 215
  Southern Hemisphere 10 | 10 | 9 | 19
Moderate renal impairment [Number; unit: participants]
  Impaired | 10 | 11 | 21
  Not impaired | 103 | 105 | 208
  Missing | 4 | 1 | 5
Screening serum albumin [Number; unit: participants] — Grade 3 (severe) = albumin < 2.0 g/dL
  Other Grade = Grades 1 (mild; 3.0 g/dL) or 2 (moderate; 2.0 - 2.9 g/dL)
  DAIDS = Division of AIDS
  participants
    Grade 3 | 6 | 8 | 14
    Other Grade | 105 | 103 | 208
    Missing | 6 | 6 | 12
Screening lymphocytes [Number; unit: participants] — Grade 3 = 350 - 499/mm^3 (severe)
  Grade 4 = < 350/mm^3 (potentially life-threatening)
  Other Grade = Grade 1 (mild; 600 - 650/mm^3) or Grade 2 (moderate; 500 - 599/mm^3)
  participants
    Grade 3/4 | 15 | 22 | 37
    Other Grade | 89 | 89 | 178
    Missing | 13 | 6 | 19
Screening neutrophils [Number; unit: participants] — Grade 3 = 500 - 749/mm^3 (severe)
  Grade 4 = < 500/mm^3 (potentially life-threatening)
  Other Grade = Grade 1 (mild; 1,000 - 1,300/mm^3) or Grade 2 (moderate; 750 - 999/mm^3)
  participants
    Grade 3/4 | 0 | 3 | 3
    Other Grade | 104 | 108 | 212
    Missing | 13 | 6 | 19
Supplemental oxygen required at Screening [Number; unit: participants]
  Yes | 75 | 83 | 158
  No | 41 | 32 | 73
  Missing | 1 | 2 | 3
Subjects who received antivirals prior to treatment [Number; unit: participants] | 88 | 82 | 170
Duration of hospital admission prior to first dose [Mean (Standard Deviation); unit: days] | 1.1 (0.98) | 1.3 (2.86) | 1.2 (2.13)
Corticosteroid at enrollment [Number; unit: participants]
  Yes | 52 | 68 | 120
  No | 65 | 49 | 114

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Influenza Virus Titer (48 Hours)
Description: The time-weighted change from baseline in log10 tissue culture infective dose50 (TCID50/mL) was calculated on a by-subject basis through 48 hours using the trapezoidal rule with all available data minus the baseline value. Ninety-five percent confidence intervals about the median time-weighted change from baseline were presented for each treatment group.
Time Frame: Baseline and 48 hours
Population: The Intent-to-Treat Infected (ITTI) population included all randomized subjects who received at least 1 dose/infusion of study drug, and had confirmed influenza A or B by culture, PCR, or serology. Overall, 83 subjects were excluded due to negative Baseline titers (log10 TCID50 0.5).
Measure: Median (95% Confidence Interval); unit: log10 TCID50/mL
Groups:
- Peramivir 300 mg: 300 mg twice daily
  Peramivir: 300 mg twice daily
- Peramivir 600 mg: 600 mg once daily
  Peramivir: 600 mg once daily
Arm/Group | Peramivir 300 mg | Peramivir 600 mg
Number analyzed (Participants) | 20 | 24
log10 TCID50/mL | -1.66 [-2.32 to -0.61] | -1.47 [-1.89 to -0.75]

2. Secondary Outcome: Change in Influenza Virus Titer, as Measured by Quantitative RT-PCR (log10 vp/mL)
Description: The time-weighted change from baseline in viral titer measured by RT-PCR was calculated on a by-subject basis through 216 hours using the trapezoidal rule with all available data minus the baseline value. Ninety-five percent confidence intervals about the median time-weighted change from baseline were presented for each treatment group.
Time Frame: Baseline, 48, 108, 216 hours
Population: The Intent-to-Treat Infected (ITTI) population included all randomized subjects who received at least 1 dose/infusion of study drug, and had confirmed influenza A or B by culture, PCR, or serology. Overall, 41 subjects were excluded due to negative Baseline titers (viral particles/mL RT-PCR value 1.58 for Influenza A and 1.49 for Influenza B).
Measure: Median (95% Confidence Interval); unit: log10 viral particles/mL
Arm/Group | Peramivir 300 mg | Peramivir 600 mg
Number analyzed (Participants) | 37 | 49
log10 viral particles/mL
  Change from baseline, 48 hours | -1.00 [-1.52 to -0.77] | -1.07 [-1.24 to -0.67]
  Change from baseline, 108 hours | -1.65 [-1.99 to -1.45] | -1.59 [-1.86 to -1.24]
  Change from baseline, 216 hours | -2.15 [-2.38 to -1.96] | -1.79 [-2.11 to -1.35]

3. Secondary Outcome: Time to Clinical Resolution
Description: Time to clinical resolution was the number of hours from initiation of study treatment until 4 of the 5 signs of clinical stability (including both body temperature and transcutaneous oxygen saturation) met resolution criteria that was maintained for at least 24 hours. The median time to clinical resolution and associated 95% confidence interval were estimated for each treatment group using the method of Kaplan-Meier. Subjects who did not achieve clinical resolution were censored at the time of their last assessment.
Time Frame: 28 days
Population: The Intent-to-Treat Infected (ITTI) population included all randomized subjects who received at least 1 dose/infusion of study drug, and had confirmed influenza A or B by culture, PCR, or serology.
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Peramivir 300 mg | Peramivir 600 mg
Number analyzed (Participants) | 56 | 70
hours | 44.7 [40.7 to 118.5] | 166.1 [84.0 to 273.1]

4. Secondary Outcome: Number of Participants With Clinical Resolution
Description: Clinical resolution was defined as normalization of at least 4 of the 5 signs of clinical stability (including both body temperature and transcutaneous oxygen saturation) for at least 24 hours.
Time Frame: 28 days
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Peramivir 300 mg | Peramivir 600 mg
Number analyzed (Participants) | 57 | 70
participants | 41 | 42

5. Secondary Outcome: Time to Alleviation of Symptoms
Description: Time to alleviation of symptoms, defined as the time from initiation of study drug until the start of the 24 hour period where all seven symptoms of influenza are recorded as none or mild, was estimated using the method of Kaplan-Meier (adolescents and adults). The 95% confidence interval about the median was presented. Subjects who did not experience alleviation of symptoms were censored at the time of the last non-missing symptom assessment.
Time Frame: 28 days
Population: The Intent-to-Treat Infected (ITTI) population included all randomized subjects who received at least 1 dose/infusion of study drug, and had confirmed influenza A or B by culture, PCR, or serology. Symptom data for 18 subjects was missing.
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Peramivir 300 mg | Peramivir 600 mg
Number analyzed (Participants) | 51 | 58
hours | 135 [89 to 184] | 158 [103 to 306]

6. Secondary Outcome: Time to Resolution of Fever
Description: Time to resolution of fever was the number of hours from initiation of study treatment until temperature was ≤37.2°C/≤99°F oral or ≤37.8°C/≤100°F rectal or tympanic for at least 24 hours with no antipyretic medication taken within 4 hours prior to the temperature measurement. Subjects who did not achieve resolution of fever were censored at the time of their last assessment. The 95% confidence interval about the median were presented.
Time Frame: 28 days
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Peramivir 300 mg | Peramivir 600 mg
Number analyzed (Participants) | 57 | 70
hours | 27.2 [12.5 to 37.0] | 24.2 [12.8 to 54.0]

7. Secondary Outcome: Time to Resumption of Usual Activities
Description: Subject's ability to perform usual activities as determined from the visual analog scale (scale ranges from 0 to 10 where 0 indicates subject was unable to perform usual activities at all and 10 indicates subject is able to perform all usual activities fully) was summarized by study visit day and treatment group. The median time to resumption of usual daily activities and associated 95% CI was estimated using the method of Kaplan-Meier for adults and adolescents. Subjects who did not return to the pre-study level of performance of usual daily activities were censored at the time of their last non-missing visual analog scale value. A separate analysis was conducted for children.
Time Frame: 28 days
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Peramivir 300 mg | Peramivir 600 mg
Number analyzed (Participants) | 53 | 59
hours | 27.7 [17.8 to NA] — The number of observed events was too small to allow estimation of the required parameter. | 24.9 [13.5 to 28.8]

8. Secondary Outcome: Time to Hospital Discharge
Description: Time to hospital discharge, defined as the number of days from initiation of study drug until the subject is discharged from the hospital, was estimated using the method of Kaplan-Meier. The 95% confidence interval about the median was presented. Subjects who were not discharged during the study period were censored at the last study visit. Subjects who died prior to discharge were censored at the longest observed time to discharge.
Time Frame: 28 days
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Peramivir 300 mg | Peramivir 600 mg
Number analyzed (Participants) | 57 | 70
days | 6 [5 to 8] | 6 [6 to 11]

9. Secondary Outcome: Number of Participants Experiencing Influenza-related Complications
Description: Influenza-related complications were defined as the occurrence of sinusitis, otitis, bronchitis and pneumonia as reported on the Influenza-related complications CRF.
Time Frame: 28 days
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Peramivir 300 mg | Peramivir 600 mg
Number analyzed (Participants) | 57 | 70
participants | 39 | 48

10. Secondary Outcome: Number of Participants Admitted to ICU After Initiation of Treatment
Description: The number of subjects experiencing ICU admission after initiation of treatment.
Time Frame: 28 days
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Peramivir 300 mg | Peramivir 600 mg
Number analyzed (Participants) | 57 | 70
participants | 2 | 6

11. Secondary Outcome: Duration of Postbaseline ICU Admission (Kaplan-Meier Estimate)
Description: The duration of ICU admission after initiation of treatment was estimated by the method of Kaplan-Meier. Subjects who were not discharged from the ICU were censored at the time of their last assessment
Time Frame: 28 days
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Peramivir 300 mg | Peramivir 600 mg
Number analyzed (Participants) | 57 | 70
days | 7 [2 to 11] | 7 [4 to 9]

12. Other Pre Specified Outcome: Number of Participants Who Required More Than 5 Days of Peramivir Treatment
Description: The number of subjects who continued more than 5 days were as reported on the Continuation of Treatment CRF page.
Time Frame: 28 days
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Peramivir 300 mg | Peramivir 600 mg
Number analyzed (Participants) | 57 | 70
participants | 16 | 28

13. Secondary Outcome: Survival (Kaplan-Meier Estimates)
Description: Survival was calculated as the number of days from initiation of study drug until death or last contact. Overall survival was estimated by the method of Kaplan-Meier; 95% confidence intervals for 14- and 28-day survival were presented by treatment group. Subjects who had not died were censored at the date of last contact.
Time Frame: 14 and 28 days
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percent Survival
Arm/Group | Peramivir 300 mg | Peramivir 600 mg
Number analyzed (Participants) | 57 | 70
Percent Survival
  14 Day Survival | 98 [88 to 100] | 93 [83 to 97]
  28 Day Survival | 94 [83 to 98] | 86 [75 to 93]

ADVERSE EVENTS:
Time Frame: Reports of AEs were collected from the time of study drug administration through the follow-up period ending on Day 14 or Day 28.
Description: For subjects who experienced the same coded event more than once, only one event is presented.
  Four of 234 randomized subjects did not receive treatment; safety analyses included 230 subjects (114 in the Peramivir 300 mg arm and 116 in the Peramivir 600 mg arm).
Arm/Group | Peramivir 300 mg | Peramivir 600 mg
Serious Adverse Events (participants affected / at risk) | 21/114 | 26/116
Other Adverse Events (participants affected / at risk) | 69/114 | 65/116
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Peramivir 300 mg (N=114) | Peramivir 600 mg (N=116)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Septic shock (Infections and infestations) | 1 | 3
Sepsis (Infections and infestations) | 1 | 2
Pneumonia bacterial (Infections and infestations) | 2 | 0
Pneumonia staphylococcal (Infections and infestations) | 2 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 3
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1
Bronchiolitis (Infections and infestations) | 1 | 0
HIV Infection (Infections and infestations) | 1 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 1 | 0
Meningococcal Bacteraemia (Infections and infestations) | 1 | 0
Pneumonia Necrotising (Infections and infestations) | 0 | 1
Pseudomonal Bacteraemia (Infections and infestations) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Hypertensive crisis (Vascular disorders) | 0 | 1
Hypoperfusion (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Multi-organ failure (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Cystic fibrosis (Congenital, familial and genetic disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Non-Hodgkin's lymphoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Mental status changes (Psychiatric disorders) | 1 | 0
Purpura (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Peramivir 300 mg (N=114) | Peramivir 600 mg (N=116)
Constipation (Gastrointestinal disorders) | 19 | 11
Diarrhoea (Gastrointestinal disorders) | 12 | 16
Nausea (Gastrointestinal disorders) | 10 | 8
Vomiting (Gastrointestinal disorders) | 4 | 4
Abdominal Distension (Gastrointestinal disorders) | 0 | 5
Gastrointestinal Sounds Abnormal (Gastrointestinal disorders) | 0 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 8 | 14
Hyperglycaemia (Metabolism and nutrition disorders) | 7 | 7
Hypophosphataemia (Metabolism and nutrition disorders) | 5 | 4
Fluid Overload (Metabolism and nutrition disorders) | 3 | 4
Hypocalcaemia (Metabolism and nutrition disorders) | 4 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 | 4
Metabolic Alkalosis (Metabolism and nutrition disorders) | 2 | 5
Hyperkalaemia (Metabolism and nutrition disorders) | 3 | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 3
Oedema Peripheral (General disorders) | 10 | 8
Oedema (General disorders) | 2 | 6
Generalised Oedema (General disorders) | 3 | 2
Pain (General disorders) | 3 | 1
Catheter Related Complication (General disorders) | 3 | 0
Insomnia (Psychiatric disorders) | 13 | 4
Agitation (Psychiatric disorders) | 2 | 6
Anxiety (Psychiatric disorders) | 5 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 5
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Respiratory Alkalosis (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Hypotension (Vascular disorders) | 7 | 11
Hypertension (Vascular disorders) | 5 | 8
Anaemia (Blood and lymphatic system disorders) | 5 | 13
Leukocytosis (Blood and lymphatic system disorders) | 4 | 4
Thrombocytosis (Blood and lymphatic system disorders) | 1 | 4
Headache (Nervous system disorders) | 7 | 5
Dizziness (Nervous system disorders) | 4 | 0
Migraine (Nervous system disorders) | 0 | 3
Urinary Tract Infection (Infections and infestations) | 5 | 2
Fungal Skin Infection (Infections and infestations) | 3 | 2
Oral Herpes (Infections and infestations) | 3 | 2
Alanine Aminotransferase Increased (Investigations) | 4 | 2
Blood Triglycerides Increased (Investigations) | 2 | 4
Aspartate Aminotransferase Increased (Investigations) | 3 | 2
Blood Potassium Decreased (Investigations) | 4 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 3
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 3 | 2
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Rash (Skin and subcutaneous tissue disorders) | 3 | 5
Erythema (Skin and subcutaneous tissue disorders) | 1 | 3
Atrial Fibrillation (Cardiac disorders) | 3 | 2
Cardiac Failure Congestive (Cardiac disorders) | 2 | 3
Renal Failure Acute (Renal and urinary disorders) | 0 | 4
Haematuria (Renal and urinary disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No